CLINICAL TRIAL: NCT06693024
Title: A Cohort Study of Adjuvant Therapy With Naratinib in HER2 Positive Early Breast Cancer
Brief Title: Adjuvant Therapy With Neratinib in HER2 Positive Early Breast Cancer
Acronym: NeraHER2
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z168
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: adjuvant therapy; neratinib
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor paraffin sample for each patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neratinib: After standard anti-HER2 neoadjuvant/adjuvant therapy, sequential targeted therapy with neratinib for 1 year
  Interventions: Drug: neratinib
- control group: After standard anti-HER2 neoadjuvant/adjuvant therapy, no sequential targeted therapy

INTERVENTIONS:
Drug: neratinib — neratinib 240mg qd for 1 year
  Groups: neratinib

SUMMARY:
Human epidermal growth factor receptor 2 (HER2) positive breast cancer is a molecular subtype with high malignancy and high risk to recurrence and metastasis. After the appearance of anti-HER2 targeted drugs, the prognosis and survival of these patients were greatly improved. In addition to trastuzumab and pertuzumab, the use of tyrosine kinase inhibitor (TKI) can further improve the survival. The evidence of previous adjuvant TKI anti-HER2 therapy was mainly from ExteNET study. However, due to the limitations of the times, ExteNET research is based on the background of only trastuzumab targeted therapy. Nowadays, there is no evidence that trastuzumab combined patuzumab,use of T-DM1, followed by sequential neratinib can still obtain absolute benefits. Therefore, there is no standard for the use of neratinib in current clinical practice. Investigators want to explore, in the real world, the efficacy and safety of sequential use of naratinib in adjuvant therapy.

DETAILED DESCRIPTION:
Investigators retrospectively recuited patients with early HER2 positive breast cancer treated in Peking University People's Hospital center from January 1, 2019 to November 31, 2024, and prospectively recruit same patients from December 1, 2024 to December 31, 2028. To compare the efficacy and safety of sequential use of neratinib.

Inclusion Criteria:

1. Patients with HER2 positive breast cancer who were diagnosed by core needle biopsy/operation in Peking University People's hospital;
2. The patients were treated in Peking University People's Hospital and underwent radical resection with hospitalization records;
3. Received standard anti-HER2 neoadjuvant/adjuvant therapy (trastuzumab, trastuzumab combined with pertuzumab, T-DM1)
4. Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

1. Lack of clinical and pathological data (such as imaging data and pathological data);
2. Patients with metastatic breast cancer or bilateral breast cancer;
3. Failure to perform radical surgery

patients recieved Neratinib for 1 year or not.

Primary end point: 5-year invasive dieased free survival

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with HER2 positive breast cancer who were diagnosed by core needle biopsy/operation in Peking University People's hospital;
* 2) The patients were treated in our hospital and underwent radical resection with hospitalization records;
* 3) Received standard anti-HER2 neoadjuvant/adjuvant therapy (trastuzumab, trastuzumab combined with pertuzumab, T-DM1)
* 4) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Patients with metastatic breast cancer or bilateral breast cancer;
* 3) Failure to perform radical surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early stage HER2 positive breast cancer patients received radical surgery and standard neoadjuvant/adjuvant therapy
Sampling Method: Probability Sample
Enrollment: 2806 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.

SECONDARY OUTCOMES:
disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
distant disease free survival | 5 years
  Time from study enrollment to distant recurrence and metastasis
breast cancer specific survival | 5 years
  Time from study enrollment to death due to breast cancer
overall survival | 5 years
  Time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China